CLINICAL TRIAL: NCT03427541
Title: A Multi-centre Real-world Non-interventional Observational Study to Explore Prognoses of the Patients With Non-small Cell Lung Cancer Complicated With Oligometastases
Brief Title: A Study to Explore Prognoses of NSCLC Patients Complicated With Oligometastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhang Helong, Professor, Tang-Du Hospital
Other Study IDs: WTONG05
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Chinese; non-small cell lung cancer; oligometastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with surgeries: NSCLC patients with surgeries
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Surgeries

SUMMARY:
An observational study to explore prognoses and clinical treatments of the patients with non-small cell lung cancer complicated with oligometastases

DETAILED DESCRIPTION:
A multi-centre real-world non-interventional observational study to explore prognoses and clinical treatments of the patients with non-small lung cancer complicated with oligometastases

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed patients with non-small cell lung cancer;
* Tumor metastases in one organ (no more than 3 metastases);

Exclusion Criteria:

* Patients with intrapulmonary metastases or multiple primary tumors;
* Patients with pleural dissemination or invasion of extrapulmonary organs;
* Patients with supraclavicular lymph node metastasis;
* Patients with systematic diseases that would influence patient survivals;
* Patients with no records for visits;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathologically diagnosed patients with non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2014 - 2017
  Overall survival

SECONDARY OUTCOMES:
Disease-free survival | 2014 - 2017
  Disease-free survival

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No